CLINICAL TRIAL: NCT02425657
Title: Fast Track Module Based Colonoscopy Training Programme for Surgical Trainees at North Jutland Surgical Departments
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Collaborators: Nordsim (Unknown)
Responsible Party: Principal Investigator, Lasse Pedersen, MD, Ph.D.-student, Aalborg University Hospital
Other Study IDs: AalborgH1
Record Dates: First submitted 2015-04-10; First posted 2015-04-24 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Harm Reduction; Perforation During Colonoscopy; Colorectal Cancer
Keywords: Education; Training; Fast track; Colonoscopy
MeSH Terms: conditions — Harm Reduction; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Junior Doctors: Surgical trainees (PGY1, 2 and 3 - Danish equivalents: introduktionsstilling, hoveduddannelse 1, 2).
  Interventions: Behavioral: Training of junior doctors

INTERVENTIONS:
Behavioral: Training of junior doctors — Training program

SUMMARY:
Specially educated trainers will be responsible for colonoscopy training of junior doctors. The educated trainers will have attended seminars held by Valori et al.

The following fast track colonoscopy training program for junior doctors will consist of: 1) Endoscopy simulation training and theory course 2) supervised and partly supervised lower endoscopy. 3) Directly observed practical skills according graded by MCSAT (Mayo Clinical Skills Assessment Tool) .

DETAILED DESCRIPTION:
Initially a "train the trainers" program will begin with 3 sessions held by Valori et al. at Aalborg University Hospital. 6 Trainers are expected to be trained during the "train the trainers" program. The doctors selected for the "train the trainers" program are doctors specialized in abdominal surgery with an extensive lower GI-endoscopy experience and who is considered to have an excellent teaching ability to educate junior doctor.

The training program for junior doctors consist of the following:

* Initial 1 day endoscopy simulation and theory at Nordsim. Endoscopy simulation scores will be monitored.
* 20 days of fully supervised colonoscopies (max booking of 6 colonoscopies pr day). Trainer is always present in the endoscopy room
* MCSAT (Mayo Clinical Skills Assessment Tool) will be used to grade the trainee multiple times and planned at day 0,5,10,15 and 20. Multiple graders will be used.
* Simulator test will be held at day 0, 10 and 20 colonoscopies to validate progress and compare simulator generated measures with MCSAT. Both the AccuTouch and Symbionix simulator will be used,

ELIGIBILITY:
Inclusion Criteria:

* Doctors currently enrolled in PGY1, 2 and 3 - Danish equivalents: introduktionsstilling, hoveduddannelse 1, 2.
* Able to arrange colonoscopy training in such a way that the total program can be completed in 12 weeks.
* Able to perform supervised upper endoscopy.

Exclusion Criteria:

* Less than 4 months left at current job position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Junior doctors in North Jutland Surgical Departments defined as PGY1, 2 and 3 - Danish equivalents: introduktionsstilling, hoveduddannelse 1, 2.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2016-09-14 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
MCSAT (Mayo Clinical Skills Assessment Tool) | 12 weeks
  Measured at day 0,5,10,15 and 20.

SECONDARY OUTCOMES:
Endoscopy training computer generated data - Percentage of colon visualized | 12 weeks
  Computer generated score (Simulator test performed at day 0, 10 and 20)
Endoscopy training computer generated data - Time to cecum | 12 weeks
  Computer generated score (Simulator test performed at day 0, 10 and 20)colonoscopies)
Endoscopy training computer generated data - Estimated patient pain | 12 weeks
  Computer generated score (Simulator test performed at day 0, 10 and 20)
Endoscopy training computer generated data: Percentage spent with clear view | 12 weeks
  Computer generated score (Simulator test performed at day 0, 10 and 20)
Endoscopy training computer generated data - Total score | 12 weeks
  Computer generated score (Simulator test performed at day 0, 10 and 20)

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Pedersen, m.d., Principal Investigator — Aaborg University Surgical Department
Locations (3):
- Denmark (3):
  - Aalborg University Hospital:Hobro, Hobro, Jutland
  - NordSim, Aalborg University Hospital, Aalborg
  - Hjörring Hospial, Hjørring

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fried GM, Marks JM, Mellinger JD, Trus TL, Vassiliou MC, Dunkin BJ. ASGE's assessment of competency in endoscopy evaluation tools for colonoscopy and EGD. Gastrointest Endosc. 2014 Aug;80(2):366-7. doi: 10.1016/j.gie.2014.03.019. No abstract available. PMID 25034851
- [Background] Preisler L, Svendsen MBS, Nerup N, Svendsen LB, Konge L. Simulation-based training for colonoscopy: establishing criteria for competency. Medicine (Baltimore). 2015 Jan;94(4):e440. doi: 10.1097/MD.0000000000000440. PMID 25634177
- [Background] Sedlack RE. Training to competency in colonoscopy: assessing and defining competency standards. Gastrointest Endosc. 2011 Aug;74(2):355-366.e1-2. doi: 10.1016/j.gie.2011.02.019. Epub 2011 Apr 23. PMID 21514931
- [Background] Kaminski MF, Anderson J, Valori R, Kraszewska E, Rupinski M, Pachlewski J, Wronska E, Bretthauer M, Thomas-Gibson S, Kuipers EJ, Regula J. Leadership training to improve adenoma detection rate in screening colonoscopy: a randomised trial. Gut. 2016 Apr;65(4):616-24. doi: 10.1136/gutjnl-2014-307503. Epub 2015 Feb 10. PMID 25670810